CLINICAL TRIAL: NCT03599232
Title: Impact of Formative Objective Structured Clinical Examination (OSCE) on Students' Summative Clinical Performance: A Randomized Controlled Trial
Brief Title: Impact of Formative OSCE on Students' Summative Clinical Performance
Acronym: OSCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Nazdar Ezzaddin Alkhateeb, Assistant Professor, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NAlkhateeb
Record Dates: First submitted 2018-06-24; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Objective Structured Clinical Examination; Clinical Performance
Keywords: formative assessment; objective structured clinical examination (OSCE); Iraq; impact; feedback
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: Students in the intervention group (first-arm) attended a formative-OSCE on the first day of their pediatric module to assess the competencies they gained from previous modules. The formative-OSCE design involved a blueprint development which served as a guideline for the development and face-validation of the 8 stations, which were both interactive and static.
  The formative-OSCE examiners consisted of 2 teaching staff and 11 postgraduate pediatric board trainees, who were trained by the researcher using role model and audiovisual aids. The formative-OSCE was carried out following the exact same process of the summative-OSCE. It composed of stations assessing same competencies with standardized mark sheets and feedback. Students received feedback on their performance in the formative-OSCE on the day the results were released on a one-to-one basis.
  at the end of pediatric module both groups undergo summative OSCEassessment
Who Masked: Outcomes Assessor
Masking Description: The staff who participated in the summative-OSCE(outcome assessor) were unaware of the group assignment and the two-teaching staff who participated in the intervention (Formative-OSCE) did not participate in the summative exam.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention( formative OSCE) (Active Comparator): students attended a formative objective structured clinical examination (OSCE) on the first day of their pediatric module to assess the competencies they gained from previous modules. the formative OSCE composed of 8 stations, which were both interactive and static. The interactive stations include history taking, examination, communication (counseling about breastfeeding), and procedural skills (pediatric basic life support) while non-interactive stations include data interpretation, management (linked-station) and a video-station (emergency).
  assessed at end of the module(7 weeks) through summative OSCE
  Interventions: Other: Formative objective structured clinical examination (OSCE)
- control (No Intervention): students in this group have attended pediatric module without formative OSCE and assessed at end of the module(7 weeks) through summative OSCE

INTERVENTIONS:
Other: Formative objective structured clinical examination (OSCE)
  Arms: intervention( formative OSCE)

SUMMARY:
Assessment is now seen as a learning experience. there is little literature on objective structured clinical examination role for formative assessment especially in developing world Many studies showed that formative-OSCE contributes positively to final summative examination performance though most studies address this point through the students' perception toward the formative-OSCE.

Having research that evaluates the effect of formative-OSCE introduction on a subsequent summative-OSCE in randomised controlled design may be of benefit for institutions considering the establishment of their own formative-OSCEs particularly in low resource countries.

DETAILED DESCRIPTION:
Formative assessments are systematically designed instructional interventions to assess and provide feedback on students' strengths and weaknesses in the course of teaching and learning and educational experts recommend its use in addition to summative assessment. Moreover, it is a requirement in undergraduate medical education and must be at the heart of student training not just included to satisfy accreditation requirement, yet unlike other professional training culture such as music in which feedback is expected, respected and given regularly to all learners, the investigators haven't cultivated a true feedback culture in medical education.

In a performance-based assessment, the Objective Structured Clinical Examination (OSCE) has gained importance because of its reliability and could be in a summative or formative manner to measure clinical competence. Clinical skills development requires time and practice at a rate that can accelerated by feedback to optimize experiential learning and improve future performance for which a learner should enter a reflection period during which available feedback is examined.

There are some medical schools where formative assessments are institutionalized and carried out systematically, unfortunately, this kind of assessment is not very frequent in Mediterranean countries.

Undergraduate medical education in Iraq is currently going through a transitional period. The Medical college of Hawler medical university (HMU) which provides a 6-year MBChB program, has started the process of changing its curriculum to competency-based medical education (CBME) and formative assessment is a requirement in this process. In the traditional curriculum training in pediatric is introduced in 5th year with summative assessment composed of 50% written test, 30% OSCE, 10% logbook, 10% history taking skills. Students should be competent to record case history, examine children, make a provisional diagnosis, interpret investigations and communicate with children and their families given that at the allotted time end, students present the case findings and evaluated by the faculty. However, a faculty member doesn't actively observe the students' actual performance of these skills or competencies so the purpose of formative assessment is not fully met. Use of OSCE as formative assessment can overcome this problem.

Attempts have been made in OSCE implementation for summative assessment, however, formative-OSCEs introduction and evaluation in Iraqi medical colleges is lacking. Iraqi medical schools are facing challenges in staff recruitment and adequate resource provision. The latter is one of the numerous concerns and challenges to the CBME implementation.

Many studies showed that formative-OSCE contributes positively to final summative examination performance though most studies address this point through the students' perception toward the formative-OSCE.

ELIGIBILITY:
Inclusion Criteria:

* 5th-year students of both gender

Exclusion Criteria:

* students who did not fulfill the 4th year requirements.
* absent on the day of performing formative OSCE
* did not agree to participate in formative OSCE

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2016-09-17 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-05-20 (Actual)

PRIMARY OUTCOMES:
performance in a summative OSCE test ( OSCE scores) | after 7 weeks from formative OSCE assessment
  The randomized groups of students with and without formative OSCE were compared on mean summative OSCE score they obtained at the end of pediatric module

SECONDARY OUTCOMES:
student feedback on formative OSCE | after completing the summative OSCE ( 7weeks after formative OSCE)
  measure students' agreement on Likert scale-based questionnaire(a scale used to represent people's attitudes to a topic.) regarding their experience in formative-OSCE (distributed to students of intervention group) the format of the scale was composed of 5 level likert items ( 5 indicating strongly agree where as 1 indicating strongly disagree)
  1. Strongly disagree (minimum)
  2. Disagree
  3. Neither agree nor disagree
  4. Agree
  5. Strongly agree ( maximum)
  the percentage of student who tick agree and strongly agree were summed to indicate student agreement on each statement in the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nazdar E. Alkhateeb, Master, Principal Investigator — Hawler Medical University; Ali A. Al-Dabbagh, Professor, Study Director — Hawler Medical University; Mohammed Ibrahim, MRCPCH, Study Chair — Queensland Health Service, Australia.; Namir G. Al-Tawil, Professor, Study Chair — Hawler Medical University
Locations (1):
- Hawler Medical University, Erbil, Kurdistan Region, Iraq